CLINICAL TRIAL: NCT05758766
Title: A Feasibility Study on the Use of Plant Based Omega-3-Fatty Acids (Flaxseed) to Improve Inflammation Driven Pain Outcomes in Children With Sickle Cell Anemia
Brief Title: Study on Use of Omega-3 Fatty Acids to Improve Outcomes in Individuals With Sickle Cell Disease
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Chinenye Dike, Assistant Professor of Pediatrics, Division of Pediatric Gastroenterology, Hepatology and Nutrition, University of Alabama at Birmingham
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-300010261; K23HL173704 (NIH)
Record Dates: First submitted 2023-02-14; First posted 2023-03-07 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Intervention Model Description: Participants will cross over after a while on plant-based omega-3-FA.
Who Masked: Participant, Investigator
Masking Description: Both principal investigator and participants will be blinded to arm of study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Regular diet (No Intervention): Participants will continue their regular diet.
- Plant based omega 3 Fatty Acid (Experimental): Participants ingest their regular diet supplemented with a plant-based omega-3-FA
  Interventions: Dietary Supplement: Plant-based omega-3-FA

INTERVENTIONS:
Dietary Supplement: Plant-based omega-3-FA — Plant-based omega 3 Fatty Acids
  Arms: Plant based omega 3 Fatty Acid

SUMMARY:
Sickle cell disease (SCD) is associated with significant morbidity and mortality. Pain and many adverse outcomes occurring in sickle cell disease are inflammatory driven. Recent data has shown that gut dysbiosis is present in individuals with sickle cell disease. Gut dysbiosis has been linked to inflammation in certain diseases. Omega -3-fatty acids (fish oil) has been shown to improve pain outcomes in individuals with sickle cell disease, but its acceptance is variable. The aim of this study is to determine if a plant-based omega-3-fatty acids will be more acceptable and also improve outcomes in individuals with sickle cell disease

DETAILED DESCRIPTION:
Sickle cell disease (SCD) is associated with significant morbidity and mortality. Pain and many adverse outcomes occurring in sickle cell disease are inflammatory driven. Recent data has shown that gut dysbiosis is present in individuals with sickle cell disease. Gut dysbiosis has been linked to inflammation in certain diseases. Omega -3-fatty acids (fish oil) has been shown to improve pain outcomes in individuals with sickle cell disease, but its acceptance is variable. The aim of this study is to determine if a plant-based omega-3-fatty acids will be more acceptable and also improve outcomes in individuals with sickle cell disease.

Children aged 5-18 years will be randomized to receive a diet rich in omega-3-fatty acids versus a regular diet for 12 weeks after which there will be a cross over of arms after a 4-week wash out period. We will compare outcomes (including patient reported pain outcomes and improvement in inflammation markers) while on the omega-3 fatty acid rich diet.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of sickle cell anemia HbSS or HbSB0 thal at steady state
* Age 5-18 years old

Exclusion Criteria:

* Age less than 5 years
* Age > 18 years old
* Chronic transfusion therapy
* Known to be pregnant
* Breastfeeding mothers
* Current use of antibiotics
* Use of pre or probiotic supplements
* PPI therapy
* Known allergy to FS

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-08-30 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Acute pain | 12 weeks
  Decrease in acute pain frequency measured with weekly pain diaries and acute care visits for pain
Chronic pain | 12 weeks
  Improvement in quality of life measured using a validated questionnaire

SECONDARY OUTCOMES:
Inflammation | 12 weeks
  Decrease in inflammation as measured by inflammatory markers

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available.